CLINICAL TRIAL: NCT05555836
Title: A Prospective Observational Study of the Association Between Cerebral Blood Flow Change and Cognitive Function in Older Maintenance Hemodialysis Patients
Brief Title: Association Between Cerebral Blood Flow Change and Cognitive Function in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Yang Luo, Chief, MD, PhD, Director of nephrology Affiliation, Beijing Shijitan Hospital, Capital Medical University
Other Study IDs: CFH2022-2-2081
Record Dates: First submitted 2022-09-17; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Hemodialysis; Cerebral Blood Flow; Cognitive Function; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of cognitive impairment in maintenance hemodialysis (MHD) patients is 3 to 5 times higher than that in ordinary people, so it is essential to find the associated risk factors in this population. This project intends to evaluate whether changes in cerebral blood flow during dialysis have an impact on cognitive function in middle-aged and elderly MHD patients and clarify their influence on brain imaging characteristics. MHD patients who started hemodialysis at 3 to 6 months were selected to examine the difference in middle cerebral artery flow rate before and after dialysis by transcranial Doppler ultrasound to reflect the changes in cerebral blood flow. Changes in the cognitive function scale assessment (memory, executive function, and other five cognitive domains) and brain magnetic resonance imaging examinations are planned to collect both at baseline and after a one-year follow-up. Then the investigator used the multiple linear regression method to analyze the effects of the difference in middle cerebral artery flow on the changes in cognitive function and the characteristics in brain imaging. The investigators anticipate that the characteristics of the influence of changes in cerebral blood flow on cognitive impairment in Chinese MHD patients will be elucidated in this study, which may provide crucial clinical evidence for finding preventive and intervention measures for cognitive impairment in this group of population.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 50, no gender limitation;
* End-stage renal disease, stable dialysis for 3-6 months;
* Subjects voluntarily participated in the study and signed informed consent, and were able to participate in clinical data collection, neuropsychological assessment, transcranial Doppler ultrasound (TCD), head MRI, and 1-year follow-up.

Exclusion Criteria:

* Congenital mental retardation or disturbance of consciousness, schizophrenia, or history of severe anxiety and depression (Hamilton Depression Scale score more than 17;
* Long-term alcohol or psychotropic drug dependence;
* Those who cannot complete the neuropsychological assessment due to visual impairment, hearing impairment, or limb dysfunction; less than 10 hours of dialysis per week;
* Patients with poor detection of the bilateral temporal window by TCD examination and unable to cooperate with ultrasound examination;
* Those who cannot undergo head MRI examination for various reasons.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese Maintenace Hemodialysis Patients
Sampling Method: Non-Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive function which is measured by MoCA scores changes after 1 year follow-up | This measurement is going to be completed within 1 year after the last participant enrolls
  This study is going to apply neuropsychological battery tests in MoCA assessment and evaluate the changes of MoCA scores of MHD patients after one year of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Luo, MD, PhD, Principal Investigator — Beijing Shijitan Hospital Affiliated to Capital Medical University
Locations (1):
- Beijing Shijitan Hospital affiliated to Capital Medical University, Beijing, China